CLINICAL TRIAL: NCT04353986
Title: Pharmacokinetics of Sofosbuvir and Ledipasvir in Hepatitis C Virus - Infected Adolescent Patients With Haematological Disorders
Brief Title: PK of SOF/LED in HCV - Infected Adolescents With Haematological Disorders
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Manal Hamdy El-Sayed, Professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL30114
Record Dates: First submitted 2019-07-15; First posted 2020-04-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: HCV Infection; Beta Thalassemia Major
Keywords: Hepatitis C virus; Pharmacokinetic Modeling; Pharmacokinetics; Sofosbuvir; Ledipasvir; Direct acting antivirals; Beta thalassemia major
MeSH Terms: conditions — Hepatitis C; beta-Thalassemia | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional, controlled, open-label, pharmacokinetic study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta thalassemia (Experimental): HCV infected Beta thalassemia major adolescents
  Interventions: Drug: Sofosbuvir and Ledipasvir
- Control (Active Comparator): HCV infected, otherwise healthy, sex and age matched to the thalassemia group serving as control group
  Interventions: Drug: Sofosbuvir and Ledipasvir

INTERVENTIONS:
Drug: Sofosbuvir and Ledipasvir — fixed dose tablet containing 400 mg sofosbuvir and 90 mg ledipasvir
  Other Names: SOF/LED

SUMMARY:
This is a prospective, controlled, open-label, pharmacokinetic study. This study aims at studying the PK of sofosbuvir, ledipasvir and sofosbuvir metabolite (GS-331007) in HCV infected children with hematological Disorders. to develop predictive pharmacokinetic model for the 3 moieties in the studied population.

In this study, patients in both treatment groups will receive 12 weeks of treatment with a fixed-dose combination tablet containing 400 mg of sofosbuvir and 90 mg of ledipasvir(SOF/LED) orally, once daily with food.

DETAILED DESCRIPTION:
In this study, patients in both treatment groups will receive 12 weeks of treatment with a fixed-dose combination tablet containing 400 mg of sofosbuvir and 90 mg of ledipasvir(SOF/LED) orally, once daily with food, as prescribed by the attending physician. Twelve eligible HCV-infected patients with hematological disorder and 12 matching HCV control patients without haematological disorder or comorbidities will be enrolled in the study. At baseline, careful history of the recruited patients including demographic characteristics (age, height, weight, and gender), comorbidities, medication history, familial history, social history, blood transfusion history, and baseline laboratory tests will be documented.

The baseline laboratory tests will include renal function tests (serum creatinine), liver function tests (bilirubin, albumin, AST, and ALT), international normalised ratio (INR), alpha fetoprotein (AFP), complete blood count (CBC), degree of liver fibrosis by Fibroscan,viral load by PCR and HCV genotype Follow-up will be done for all participants at baseline, after 10 days of treatment for the evaluation of the steady state PK parameters of SOF/LED in those patients, after 12 weeks of treatment, and after 12 weeks from the end of treatment. For a total of 4 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Adolescents (ages 12-18 years) and/ or weight more than 35 Kg
* Diagnosed with beta-thalassemia major and receiving regular blood transfusion
* spleenectomised
* Chronic HCV infection (defined as more than 6 months history of the disease)
* Naïve non-cirrhotic population with FIB Score: F0 to F3 as measured by Fibroscan
* Screening laboratory values of the beta-thalassemia group within the following thresholds (absolute neutrophil count > 1500/mm3, platelets > 7500 cells/mm3 , Serum creatinine < 1.2 mg/dl, creatinine clearance > 40 mL/min, albumin >3.5 gm/dl, and aspartate transaminase (AST) and alanine transaminase (ALT) level less than 5 fold of the normal limit). Control group should have normal biochemical profile.
* Assent of the patients and consent of their legal guardians are required

Exclusion Criteria:

* Previous treatment for HCV.
* History of clinically significant illness or any other medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol or affect the pharmacokinetics of the study drugs. Such as,

  * Ongoing or untreated cancer including haematologic and hepatic cancers
  * Co-infection with human immunodeficiency virus (HIV), acute hepatitis A virus or hepatitis B virus
  * Clincal hepatic decompensation (i.e., ascites, encephalopathy or variceal haemorrhage)
  * Renal dysfunction
  * Active infection (any infection showing clinical manifestation at time of sampling)
* Known hypersensitivity to study medications
* Ongoing treatment with cyclosporine, rifampin, phenytoin, carbamazepine, phenobarbital, or amiodarone.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Predictive Pharmacokinetic Model | 10 days
  serial blood samples will be withdrawn to measure the drug level develop a Predictive Pharmacokinetic Model for sofosbuvir, ledipasvir and GS 331007
sustained virologic response | 6 months
  sustained virologic response

SECONDARY OUTCOMES:
adverse drug reactions | 3 months
  record any adverse drug reactions experienced by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Manal H El-Sayed, M.D, Principal Investigator — Director of MARSI-CRC
Locations (1):
- Masri-Crc, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Baraky IA, Abbassi MM, Ebeid FS, Hassany M, Sabry NA, El-Sayed MH. Beta-thalassemia major alters sofosbuvir/ledipasvir exposure in Hepatitis C virus infected adolescent patients. Clin Res Hepatol Gastroenterol. 2021 Sep;45(5):101747. doi: 10.1016/j.clinre.2021.101747. Epub 2021 Jun 26. PMID 34186262